CLINICAL TRIAL: NCT02999074
Title: A Randomized 3-arm Exercise Intervention Trial for Breast Cancer Patients Undergoing Neoadjuvant Chemotherapy
Brief Title: Exercise Interventions for Breast Cancer Patients Undergoing Neoadjuvant Chemotherapy
Acronym: BENEFIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BENEFIT
Record Dates: First submitted 2016-05-06; First posted 2016-12-21 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: exercise; resistance training; aerobic training; breast cancer; neoadjuvant chemotherapy; fatigue; quality of life; tumor response
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resistance exercise (Active Comparator)
  Interventions: Other: Resistance exercise
- Aerobic exercise (Active Comparator)
  Interventions: Other: Aerobic exercise
- Waitlist control (Other)
  Interventions: Other: Usual care during neoadjuvant chemotherapy/Exercise after surgery

INTERVENTIONS:
Other: Resistance exercise — The training will take place twice weekly over the course of neoadjuvant CTx at the NCT Heidelberg or in regional qualified centers under supervision and guidance of experienced exercise therapists. The progressive resistance exercise comprises 8 machine-based exercises, each performed in 3 sets, 12 repetitions at 60-80% of one repetition maximum (1-RM).
  Arms: Resistance exercise
Other: Aerobic exercise — The training will take place twice weekly over the course of neoadjuvant CTx at the NCT Heidelberg or in regional qualified centers under supervision and guidance of experienced exercise therapists. The aerobic exercise will be performed on a cycle ergometer (or alternatively at a treadmill, elliptical, rowing ergometer, or combination) progressing from 60% to 70% VO2max with increasing duration. During weeks 7-18 the goal is to perform an extensive interval training.
  Arms: Aerobic exercise
Other: Usual care during neoadjuvant chemotherapy/Exercise after surgery — The control group receives no exercise intervention during neoadjuvant CTx, which reflects the usual care condition. To investigate effects of different exercise timing, and to provide those patients also a potential health benefit and reduce drop-out and contamination, the control group will receive 18 weeks resistance or aerobic exercise (according to their personal preferences) after breast cancer surgery.
  Arms: Waitlist control

SUMMARY:
The BENEFIT-Study is a randomized controlled 3-arm intervention trial investigating the currently discussed hypothesis that exercise concomitant to chemotherapy (CTx) may have a beneficial effect on cancer prognosis by boosting the anti-tumoral effect of the cytostatics or by enhancing therapy compliance. This hypothesis is based on pre-clinical and exploratory clinical trials. Breast cancer patients scheduled for neoadjuvant CTx will be randomized to either a resistance training or an aerobic training concomitant to the neoadjuvant CTx, or a waiting list control group that will get no exercise intervention during neoadjuvant CTx (i.e. usual care) but will exercise after breast surgery. The primary study endpoint is the tumor size. Further, the effects of resistance and aerobic exercise on the clinical-pathologic stage (CPS-EG) score, the pathological complete response (pCR), tolerability and compliance to CTx, physical fitness, patient reported outcomes such as fatigue, sleep problems, quality of life, depressive symptoms, anxiety and pain, as well as cognitive function, and selected biomarkers will be investigated.

A confirmation of the study hypothesis would be a strong argument for patients to engage in exercise as early as during neoadjuvant CTx. The trial will also provide evidence-based guidance for patients regarding type and timing of training.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of Age
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy
* Scheduled for neoadjuvant CTx (but not yet started)
* Confirmed hormone receptor and Her2 status
* Sufficient German language skills
* Willing to train at the exercise facilities twice per week

Exclusion Criteria:

* Any physical or mental conditions that would hamper the adherence to the training programs or the completion of the study procedures
* Engaging in systematic intense exercise training (at least 1h twice per week)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Tumor size | change from baseline (before start of neoadjuvant chemotherapy) to breast surgery
  percentage of change from the maximal diameter of the lesion assessed before neoadjuvant chemotherapy (by mammography or sonography) to the maximal diameter of the tumor assessed after neoadjuvant chemotherapy at breast surgery

SECONDARY OUTCOMES:
CPS-EG score | at breast surgery
  The Clinical-Pathologic Stage (CPS-EG) score combines clinical tumor stage prior to neoadjuvant therapy (CS), pathological tumor stage after neoadjuvant treatment (PS), estrogen receptor status (E) and grading (G). It has been shown to be a valid prognostic factor to discriminate among patient subgroups with respect to survival after neoadjuvant CTx.
pCR | at breast surgery
  The Pathological Complete Response (pCR) is defined as ypT0/is ypN0 and has been consistently demonstrated to be a good prognostic factor for long-term benefit from neoadjuvant CTx.
Fatigue Assessment Questionnaire (FAQ) | at baseline, week 9, post-chemotherapy (before breast surgery); months 6 and 12 after breast surgery
  Validated 20-item multidimensional self-assessment questionnaire to assess the physical, affective, and cognitive dimension of cancer-related fatigue
EORTC QLQ-C30 / BR23 | at baseline, week 9, post-chemotherapy (before breast surgery); months 6 and 12 after breast surgery
  Validated 30-item self-assessment questionnaire to assess quality of life aspects.
Patient Health Questionnaire for Depression and Anxiety (PHQ-4) | at baseline, week 9, post-chemotherapy (before breast surgery); months 6 and 12 after breast surgery
  A validated 4-item screener for depression and anxiety.
Pittsburgh Sleep Quality Index (PSQI) | at baseline, week 9, post-chemotherapy (before breast surgery); months 6 and 12 after breast surgery
  Validated questionnaire to assess sleep quality and sleep problems.
Spiroergometry (VO2max) | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
Isometric and isokinetic muscle strength measured by ISOMED 2000 | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
Body mass index | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
Self-developed physical activity questionnaire including type, duration, frequency and intensity of sports, cycling,and walking | Follow-up (6 months and 12 months after breast surgery)
Cognitive function - HVLT-R | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
  Hopkins Verbal Learning Test - Revised (HVLT-R)
Cognitive function - TMT | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
  Trail Making Test
Cognitive function - COWA | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
  Controlled Oral Word Association
Sleep quality | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
  Measured with ActiGraph (accelerometry)
Sleep efficiency | at baseline, post-chemotherapy (before breast surgery); month 6 after breast surgery
  Measured with ActiGraph (accelerometry)

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Tumor Diseases (NCT), Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haussmann A, Schmidt ME, Goldschmidt S, Hiensch AE, Wiskemann J, Steindorf K. Effects of aerobic or resistance exercise on sleep and cancer-related fatigue in patients with breast cancer during or after neoadjuvant chemotherapy: a 3-arm randomized controlled trial. BMC Med. 2026 Jan 28. doi: 10.1186/s12916-026-04669-3. Online ahead of print. PMID 41593692
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Goldschmidt S, Schmidt ME, Rosenberger F, Wiskemann J, Steindorf K. Patterns and influencing factors of exercise attendance of breast cancer patients during neoadjuvant chemotherapy. Support Care Cancer. 2024 Jan 3;32(1):79. doi: 10.1007/s00520-023-08269-2. PMID 38170301
- [Derived] Kreutz C, Muller J, Schmidt ME, Steindorf K. Comparison of subjectively and objectively assessed sleep problems in breast cancer patients starting neoadjuvant chemotherapy. Support Care Cancer. 2021 Feb;29(2):1015-1023. doi: 10.1007/s00520-020-05580-0. Epub 2020 Jun 19. PMID 32556623